CLINICAL TRIAL: NCT03657784
Title: Pharmacokinetics, Dialysability and Safety of P03277, a New Gadolinium-based Contrast Agent, in Healthy Volunteers and in Patients With Impaired Renal Function
Brief Title: Pharmacokinetics, Dialysability and Safety of P03277 in Healthy Volunteers and in Patients With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: GDX-44-005; 2017-001211-36 (EudraCT Number)
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-02

CONDITIONS: Renal Insufficiency; Healthy Volunteers
MeSH Terms: conditions — Renal Insufficiency | interventions — gadopiclenol

STUDY DESIGN:
Intervention Model Description: Successive cohorts design and single dose administration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): P03277 will be administered to healthy volunteers with stable normal renal function defined with an absolute value of eGFR ≥ 90 mL/min.
  Interventions: Drug: P03277
- Cohort 2 (Experimental): P03277 will be administered to patients with stable mild renal impairment defined with an absolute value of eGFR between 60 and 89 mL/min.
  Interventions: Drug: P03277
- Cohort 3 (Experimental): P03277 will be administered to patients with stable moderate renal impairment defined with an absolute value of eGFR between 30 and 59 mL/min.
  Interventions: Drug: P03277
- Cohort 4 (Experimental): P03277 will be administered to patients with stable severe renal impairment defined with an absolute value of eGFR between 15 and 29 mL/min.
  Interventions: Drug: P03277
- Cohort 5 (Experimental): P03277 will be administered to patients with end-stage renal failure who requires 3 hemodialysis sessions per week.
  Interventions: Drug: P03277

INTERVENTIONS:
Drug: P03277 — Single intravenous bolus injection at 0.1 mmol/kg body weight at a rate of 2 mL/second
  Other Names: gadopiclenol

SUMMARY:
This is an open-label, non-randomized, successive cohorts design, multicenter, single dose phase I study.

The primary objectives are:

* to evaluate the pharmacokinetics (plasma and urine) profile of P03277 following single intravenous injection (0.1 mmol/kg body weight) in patients with mild to severe renal impairment and in healthy volunteers with normal renal function used as reference.
* to assess dialysability of P03277 following a single intravenous injection (0.1 mmol/kg body weight) in patients with end stage renal disease requiring hemodialysis.

DETAILED DESCRIPTION:
A full range design including the different degrees of renal impairment and healthy volunteers used as reference has been chosen.

Enrolment will be successive starting with both healthy volunteers (cohort 1) and patients with mild renal impairment (cohort 2), then patients with moderate renal impairment (cohort 3), then patients with severe renal impairment (cohort 4) to end with patients with end stage renal disease (cohort 5). Pharmacokinetics and safety profiles following the confinement period will be reviewed per each successive cohort by a Data Monitoring Committee before starting recruitment of patients in the next cohort. Cohorts 1 and 2 will be recruited in parallel and Data Monitoring Committee review will start after the completion of these first two cohorts.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Subject being 18 years or older, able and willing to participate in the trial
* Subject in good enough health status as determined by investigator according to medical history, physical examination, vital signs, 12 lead ECG and laboratory tests at screening and inclusion

For healthy volunteers / cohort 1:

Healthy volunteer with stable normal renal function defined with an absolute value of eGFR ≥ 90 mL/min based on two eGFR assessments done at screening and inclusion, with a maximum tolerance of 15% between the 2 measurements

For patients with renal impairment / cohorts 2 to 5:

* Cohort 2: patient with stable mild renal impairment defined with an absolute value of eGFR between 60 and 89 mL/min included based on two eGFR assessments done at screening and inclusion, with a maximum tolerance of 15% between the 2 measurements
* Cohort 3: patient with stable moderate renal impairment defined with an absolute value of eGFR between 30 and 59 mL/min included based on two eGFR assessments done at screening and inclusion, with a maximum tolerance of 15% between the 2 measurements
* Cohort 4: patient with stable severe renal impairment defined with an absolute value of eGFR between 15 and 29 mL/min included based on two eGFR assessments done at screening and inclusion, with a maximum tolerance of 15% between the 2 measurements
* Cohort 5: patient with end-stage renal failure who requires 3 hemodialysis sessions per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
AUC | Prior to P03277 administration and at 2, 5, 10, 20, 30, 45 minutes and at 1, 2, 4, 6, 8, 12, 24 hours after administration for all cohorts. Additionally, after P03277 administration at 48 hours (cohorts 2-3-4), 72 hours (cohort 3) and 96 hours (cohort 4)
  AUC: area under the plasma concentration curve. Blood samples will be collected.
Cmax | Prior to P03277 administration and at 2, 5, 10, 20, 30, 45 minutes and at 1, 2, 4, 6, 8, 12, 24 hours after administration for all cohorts. Additionally, after P03277 administration at 48 hours (cohorts 2-3-4), 72 hours (cohort 3) and 96 hours (cohort 4)
  Cmax: peak concentration. Blood samples will be collected.
t1/2 | Prior to P03277 administration and at 2, 5, 10, 20, 30, 45 minutes and at 1, 2, 4, 6, 8, 12, 24 hours after administration for all cohorts. Additionally, after P03277 administration at 48 hours (cohorts 2-3-4), 72 hours (cohort 3) and 96 hours (cohort 4)
  t1/2: terminal half-life. Blood samples will be collected.
CLT | Prior to P03277 administration and at 2, 5, 10, 20, 30, 45 minutes and at 1, 2, 4, 6, 8, 12, 24 hours after administration for all cohorts. Additionally, after P03277 administration at 48 hours (cohorts 2-3-4), 72 hours (cohort 3) and 96 hours (cohort 4)
  CLT: total clearance. Blood samples will be collected.
Ae | Prior to P03277 administration and during the intervals 0-6, 6-24, 24-48 hours for all cohorts + during 48-72 and 72-96 hours intervals for cohorts 2-3-4, 96-120 hours interval for cohorts 3-4, 120-144 hours and 144-168 hours intervals for cohort 4
  Ae: amount excreted. Urine samples will be collected.
Relative amount of eliminated P03277 in blood | Just before the start of the session and at 30, 90 minutes and 4 hours after the start of the session.
  This outcome will be assessed for cohort 5 only. Venous blood samples will be collected at each session of hemodialysis.
Clearance of P03277 | Just before the start of the session and at 30 and 90 minutes after the start of the session.
  This outcome will be assessed for cohort 5 only and at the first hemodialysis only. Arterial and venous blood samples will be collected.
Dialysis clearance of P03277 | Just before the start of the session and at 30, 90 minutes and 4 hours after the start of the session.
  This outcome will be assessed for cohort 5 only. Venous blood and dialysate samples will be collected at each session of hemodialysis.

SECONDARY OUTCOMES:
P03277concentration in blood (long-term) | At 1, 3 and 6 months after P03277 administration
  Blood samples will be collected.
P03277 concentration in urine (long-term) | At 1, 3 and 6 months after P03277 administration
  Urine samples will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Penescu Mircea, MD, Principal Investigator — Arensia Phase I unit "Carol Davila" Nephrology Hospital
Locations (2):
- Republican Clinical Hospital, Arensia EM Unit, Chisinau, Moldova
- Arensia Phase I unit "Carol Davila" Nephrology Hospital, Bucharest, Romania

REFERENCES:
- [Derived] Bradu A, Penescu M, Pitrou C, Hao J, Bourrinet P. Pharmacokinetics, Dialysability, and Safety of Gadopiclenol, a New Gadolinium-Based Contrast Agent, in Patients With Impaired Renal Function. Invest Radiol. 2021 Aug 1;56(8):486-493. doi: 10.1097/RLI.0000000000000764. PMID 34197356